CLINICAL TRIAL: NCT04959565
Title: Evaluation of a Practice-oriented Recovery Program for Female Endurance Athletes With Relative Energy Deficiency - The FUEL Programme
Brief Title: Evaluation of a Practice-oriented Recovery Program for Female Endurance Athletes With Relative Energy Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monica Klungland Torstveit (Other)
Collaborators: Olympiatoppen (Unknown); Sport Ireland Institute (Unknown); Technical University of Munich (Other); Linnaeus University (Other)
Responsible Party: Sponsor-Investigator, Monica Klungland Torstveit, Professor, University of Agder
Organization: University of Agder (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: The FUEL program
Record Dates: First submitted 2021-06-23; First posted 2021-07-13 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Relative Energy Deficiency in Sport
MeSH Terms: conditions — Relative Energy Deficiency in Sport

STUDY DESIGN:
Intervention Model Description: One group will receive video lectures + individual consultations, while the other intervention group will receive video lectures only.
  A control group was planned for Spring 2020 but do to the COVID-19 pandemic the investigators had to cancel the reqruitment of the control group.
  Now the investigators plan a new recruitment of a control group for Authum 2021.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 16 online lectures in sports nutrition + 8 individual consultations for 16 weeks (Experimental): Non-smoking, non-contraceptive using, competitive female endurance athletes, 18-35 years of age, training a minimum of five times per week will be recruited through social media and endurance sports clubs (running, cycling, orienteering, triathlon, biathlon, and cross-country skiing) in Norway, Sweden, Germany, and Ireland.
  Athletes with a LEAF-Q score ≥8 + EDE-Q score < 2.5 who meets the other inclusion criteria will be invited for further participation.
  The lectures are designed for female endurance athletes at risk of RED-S. The participants will get access to a new lecture every week during the intervention.
  Interventions: Behavioral: Nutritional behavioral intervention
- Control (No Intervention): Non-smoking, non-contraceptive using, competitive female endurance athletes, 18-35 years of age, training a minimum of five times per week will be recruited through social media and endurance sports clubs (running, cycling, orienteering, triathlon, biathlon, and cross-country skiing).
  Athletes with a LEAF-Q score ≥8 + EDE-Q score < 2.5 who meets the other inclusion criteria will be invited for further participation.
- 16 online lectures in sports nutrition for 16 weeks (Experimental): Non-smoking, non-contraceptive using, competitive female endurance athletes, 18-35 years of age, training a minimum of five times per week will be recruited through social media and endurance sports clubs (running, cycling, orienteering, triathlon, biathlon, and cross-country skiing) in Norway, Sweden, Germany, and Ireland.
  Athletes with a LEAF-Q score ≥8 + EDE-Q score < 2.5 who meets the other inclusion criteria will be invited for further participation.
  The lectures are designed for female endurance athletes at risk of RED-S. The participants will get access to a new lecture every week during the intervention.
  Interventions: Behavioral: Nutritional behavioral intervention

INTERVENTIONS:
Behavioral: Nutritional behavioral intervention — The participants will get access to an online platform where the FUEL recovery program will be initiated with session 1 immediately after baseline testing and the athletes are requested to follow the lectures lead by highly experienced sports dietitians for the respective weeks. Every other week for 16 weeks (8 sessions in total) participants will be offered individual nutrition counselling (one intervention group) by highly experienced sports nutritionists in each country, based on Motivational Interviewing, the individual's environmental and biological prerequisites, and the Transtheoretical Model, focusing on the individual's readiness to act on a new healthier behavior
  Arms: 16 online lectures in sports nutrition + 8 individual consultations for 16 weeks
Behavioral: Nutritional behavioral intervention — The participants will get access to an online platform where the FUEL recovery program will be initiated with session 1 immediately after baseline testing and the athletes are requested to follow the lectures lead by highly experienced sports dietitians for the respective weeks.
  Arms: 16 online lectures in sports nutrition for 16 weeks

SUMMARY:
The aim of this study is to develop, implement and evaluate the effects of a 16 week practice orientated sports nutrition education and counselling program aiming to improve energy availability and to investigate the effects on physiological and psychological health, sports nutrition knowledge, and athletic performance in well-trained female endurance athletes with risk of RED-S. The FUEL (in Norwegian: Forstå Utholdenhetsidretts Ernæring - et Læringsprogram; in English: Food and nUtrition for Endurance athletes - a Learning program) recovery program consists of virtual lectures with central themes within sports nutrition in addition to individual consultations.

DETAILED DESCRIPTION:
The current project is a reversed version of the original project which included a wide range of laboratory measurements, but due to the COVID-19 pandemic the investigators had to change the test protocol to a "corona friendly" version without any physical contact between the investigators and the participants. The cancellation of laboratory tests affects many key aspects and outcomes of the project's initial plan, including the initial primary outcome energy availability which require accurate measurement of fat free mass. This ungoing project is therefore marked by the drastic decisions that had to be made immediately before recruitment considering the corona pandemic.

The investigators aim to develop, implement and evaluate a 16-week practice orientated online sports nutrition education and counselling program for female endurance athletes at risk of RED-S. The study will be evaluated in terms of changes in self-reported physiological and psychological health parameters as well as the participants' reported experiences.

A systematic evaluation of the FUEL program will be provided based on the RE-AIM framework.

The following research questions will be addressed:

Can the FUEL recovery program...

* reduce LEAF-Q score in female endurance athletes with risk of RED-S?
* improve reproductive function in female endurance athletes with MD?
* reduce EDE-Q and DT score in female endurance athletes with risk of RED-S?
* improve quality of life in female endurance athletes with risk of RED-S?
* improve sports nutrition knowledge in female endurance athletes with risk of RED-S?
* improve performance in female endurance athletes with risk of RED-S?
* improve sports nutrition habits in female endurance athletes with risk of RED-S?
* improve carbohydrat availability in female endurance athletes with risk of RED-S?
* reduce EAI score in female endurance athletes with risk of RED-S?
* recover menstrual function in female endurance athletes with MD assessed 6- or 12-months post intervention?

Additional research questions are:

* How do the participants experience to be part of the FUEL recovery program?
* How do the nutritional counselors experience the feasibility of the FUEL recovery program?
* How feasible is the FUEL program based on the RE-AIM framework?

Participants will be included in their athleic off-season and data will be conducted at baseline and at week 17 (immediately after the 4-month intervention). For the qualitative part of the FUEL project (interviews about participant experiences), data will be conducted approximately 1 month after end intervention.

An information letter will be available at the FUEL homepage (www.uia.no/fuel), and a link to the part 1 (screening) questionnaire will be available about two months before baseline testing (part 2). For the screening phase (part 1) volunteers will be asked to complete the Eating Disorder Examination Questionnaire (EDE-Q), the LEAF-Q, and the Exercise Addiction Inventory (EAI) besides additional background information (e.g. educational level). Athletes with a LEAF-Q score ≥8, will be invited to participate in the intervention (part 3) initiating with a baseline data collection week (part 2) and ending with a post intervention data collection week (part 4). Athletes with a global EDE-Q score ≥ 2.5 will be excluded due to high risk of EDs and thus high risk of non-compliance to this intervention. Part 2 and 4 includes a seven-day prospective weighed diet and activity record, an online questionnaire with questions concerning athletic performance, sports nutrition habits, self-efficiacy, drive for thinness, and quality of life as well as a welcome telephone call, including twenty statements about sports nutrition for endurance athletes.

Follow-up will be conducted 6 and 12 months post intervention.

Randomization of participants within the same geographical research site is considered unreasonable due to the high risk of imitation of intervention. Therefore, the investigators plan a waitlist control group starting with a 16-week period, including testing and questionnaires without the FUEL recovery program followed by the 16-week FUEL intervention.

The virtual lectures will be based on sports nutrition recommendations for female endurance athletes according to international peer reviewed consensus statements. The participants will get access to an online platform where the FUEL recovery program will be initiated with session 1 the week after baseline testing and the athletes are requested to follow the lectures lead by highly experienced sports dietitians for the respective weeks. Every other week for 16 weeks (8 sessions in total) participants will be offered individual nutrition counselling by highly experienced sports nutritionists in each country, based on Motivational Interviewing, the individual's environmental and biological prerequisites, and the Transtheoretical Model, focusing on the individual's readiness to act on a new healthier behavior.

In order to evaluate the FUEL recovery program based on the RE-AIM framework, an evaluation questionnaire as well as qualitative interviews will be performed post intervention for athletes and their nutrition counsellors.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Non-contraceptive using
* Competitive female endurance athletes
* 18-35 years of age
* training minimum 5 times a week
* Athletes with LEAF-Q score ≥ 8 and EDE-Q score < 2.5 from part 1 will be invited to participate in the 16 week FUEL intervention

Exclusion Criteria:

* Pregnancy or planned pregnancy
* Risk of eating disorders defined as an EDE-Q score ≥ 2.5
* chronic diseases (e.g. diabetes, crohn's disease, thyroid dysfunction)
* Use of any medication that may disturb hormonal balance

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females as innate sex
Enrollment: 50 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Low Energy Availability in Females Questionnaire score | 16 weeks
  In this reversed project description, the primary outcome will be change in LEAF-Q score from pre- to post intervention.
  Low Energy Availability in Females Questionnaire (LEAF-Q) assess menstrual funktion, gatsrointestinal funktion and injuries and have been widely used to detect female athletes at risk for RED-S. The questinnaire have been validated in Scandinavian female elite endurance athletes. A score of 8 or more is assessed as a sign of low energy availability.
  Based on an initial analysis during the recruitment phase with an expected improvement in LEAF-Q score of 3 and Type I and Type II error of 5% and 20% respectively, the power calculation suggest 28 subjects in each group. To account for dropouts, the investigators aim for 35 participants in each group.

SECONDARY OUTCOMES:
Menstrual bleeding frequency | 16 weeks
  Self-reported using BESTR
Eating Disorder examination questionnaire (EDE-Q 6.0) | 16 weeks, 6 and 12 months
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-reported questionnaire adapted from the semi-structured interview Eating Disorder Examination. Each question can be answered on a scale from 0 to 6. Higher score means higher risk of eating disorder.
  It is designed to assess the range and severity of features associated with a diagnosis of eating disorder using 4 subscales (Restraint, Eating Concern, Shape Concern and Weight Concern) and a global score.
Quality of Life (WHOQOL-BREF) | 16 weeks, 6 and 12 months
  World Health Organization Quality of Life-BREF (WHOQOL-BREF). Each answer will be converted to a point from 1-5 by the scienists, where higher score equals better quality of life.
Self-perceived knowledge about sports nutrition | 16 weeks, 6 and 12 months
  Five self-constructed questions which is rank on a scale from 1 to 10. Higher score means higher self-perceived knowledge about sports nutrition.
Sport performance | 16 weeks, 6 and 12 months
  Ten self-constructed questions in relation to the RED-S model concerning self-experienced athletic performance the last 4 weeks. Each question will be answered on a scale from 1-10 with alternating "good" or "bad" performance for high and low values, respectively.
Participant evaluation | 1 week after end intervention
  An online questionnaire containing 21 questions regarding the participants' evaluation of the FUEL intervention. The questionnaire contains both open and closed questions. Questions with answers on a scale from 1 to 10 will be presented as mean +/- SD, while others will be presented as a percentage or in text (for open questions).
Sports nutrition related behavior | 16 weeks, 6 and 12 months
  Eight self-constructed questions regarding sports nutrition behavior the last 4 weeks. All questions are closed with different frequency categories. These will be presented as a percentage.
Experiences with participation in the FUEL project | Approximately four weeks after end intervention
  Qualitative interviews with participants and their nutrition supervisors. An interview guide will be followed for the participants and the supervisors, respectively. An investigator who has not been a part of the development or the implementation of the FUEL intervention itself, will be conducting the interviews.
Exercise addiction | 16 weeks, 6 and 12 months
  The exercise addiction inventory (EAI) is a short screening tool consisting of six questions based upon the six components of addiction. Each question can be answered on a scale from 1-5. Higher score means higher risk of exercise addiction.
Eating Disorder Inventory (EDI) subscale score Drive for Thinness (DT) | 16 weeks, 6 and 12 months
  EDI DT score have previously been found as a proxy indicator of energy deficiency in exercising women. The DT scale consist of seven questions about attitudes and behaviors concerning eating, weight, and shape. Each question has six possible answers which corresponds to a score from 0 to 4. Higher score means higher drive for thinness.
Knowledge about sports nutrition for female endurance athletes | 16 weeks
  A telephone interview where the investigator reads out 20 claims about sports nutrition. The participant has the possibility to answer "true", "false" or "unsure". A higher percentage of correct answer means better knowledge about sports nutrition.
Appetite | 16 weeks
  Every day during the baseline testing week, during the intervention and during the post intervention week, participants are encouraged to rank their level of appetite in BESTR training diary on a scale from 1 to 10, 1 corresponding to no appetite and 10 corresponding to a great degree of appetite.
Readiness to train | 16 weeks
  Every day during the baseline testing week, during the intervention and during the post intervention week, participants are encouraged to rank their level of readiness to train in BESTR training diary on a scale from 1 to 10, 1 corresponding to not ready at all and 10 corresponding to a great degree of readiness to train.
Sleep quality | 16 weeks
  Every day during the baseline testing week, during the intervention and during the post intervention week, participants are encouraged to rank their sleep quality in BESTR training diary on a scale from 1 to 10, 1 corresponding to low and 10 corresponding to a high sleep quality.
Sleep quantity | 16 weeks
  Every day during the baseline testing week, during the intervention and during the post intervention week, participants are encouraged their daily sleep in hours and minutes in BESTR training diary.
Carbohydrate availability | 16 weeks
  Participants are ask to register all foods and beverages during the baseline registration week and the post intervention week. Carbohydrate availability will be expressed in g/kg body weight and compared to current sports nutrition guidelines.
Nutrients | 16 weeks
  Participants are ask to register all foods and beverages during the baseline registration week and the post intervention week. Nutrients will be analyzed in Dietist Net for Norwegian and Swedish athletes, Nutritics for Irish athletes, and EBISpro for German athletes.

CONTACTS AND LOCATIONS:
Overall Officials: Monica K Tortsveit, Professor, Study Director — University of Agder
Locations (4):
- Technical University of Munich, Munich, Germany
- Sport Ireland Institue, Dublin, Ireland
- University of Agder, Kristiansand, Norway
- Linnaeus University, Kalmar, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fahrenholtz IL, Melin AK, Garthe I, Wasserfurth P, Ivarsson A, Hollekim-Strand SM, Koehler K, Logue D, Madigan S, Grafnings M, Torstveit MK. Short-term effects and long-term changes of FUEL-a digital sports nutrition intervention on REDs related symptoms in female athletes. Front Sports Act Living. 2023 Dec 18;5:1254210. doi: 10.3389/fspor.2023.1254210. eCollection 2023. PMID 38164441